CLINICAL TRIAL: NCT00334321
Title: Pelvic IMRT With Tomotherapy: A Phase I Feasibility Study in Post-Hysterectomy Endometrial Cancer Patients
Brief Title: Pelvic IMRT With Tomotherapy in Post-Hysterectomy Endometrial Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0297 / 201106410
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Endometrial Cancer
Keywords: IMRT; Tomotherapy; Post-Hysterectomy; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMRT with chemotherapy (Experimental): IMRT (upper third of vagina & para-vaginal tissue and the common, external and internal iliac nodal regions) 160-180 cGy daily fractions for a total dose of 4500-5120 cGy. Once a day treatment four to five days a week for approximately 6 weeks.
  Intracavitary vaginal brachytherapy - some patients will be given this and it will be decided by the treating physician.
  Carboplatin - AUC 6, IV over 30-60 minutes following completion of paclitaxel, given once every 3 weeks (3 weeks=1 cycles) for a total of 6 cycles
  Paclitaxel - 175 mg/m2, 3 hour continuous IV infusion, administered prior to carboplatin, given once every 3 weeks (3 weeks=1 cycles) for a total of 6 cycles
  Interventions: Radiation: IMRT; Radiation: Intracavitary vaginal brachytherapy; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: IMRT
Radiation: Intracavitary vaginal brachytherapy
Drug: Paclitaxel
  Other Names: Taxol
Drug: Carboplatin

SUMMARY:
This study is evaluating the feasibility of using helical tomotherapy to deliver IMRT in post-hysterectomy endometrial cancer patients receiving adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years of age
2. Karnofsky Performance Status of greater than or equal to 60
3. FIGO Surgical Stage I, II, and III
4. Pathologic confirmation of endometrial cancer
5. Patient status post hysterectomy
6. Patients with local or regional metastases are eligible for this protocol, but not those with distant metastases
7. Patients must have adequate:

   * Bone Marrow Function:

     * ANC ≥ 1,500/mcl (< CTCAE v 3.0 Grade 1).
     * Platelets ≥ 100,000/mcl (< CTCAE v3.0 Grade 1).
   * Renal Function:

     * Serum creatinine ≤ institutional upper limit normal (ULN) (CTCAE v 3.0 Grade 0). Note: if serum creatinine > ULN, a 24-hour creatinine clearance must be collected and must be > 50 mL/min.
   * Hepatic Function:

     * Bilirubin ≤ 1.5 x ULN (< CTCAE v 3.0 Grade 1).
     * SGOT≤ 2.5 x ULN (< CTCAE v 3.0 Grade 1).
     * Alkaline phosphatase ≤ 2.5 x ULN (< CTCAE v 3.0 Grade 1).
   * Neurologic Function:

     * Neuropathy (sensory and motor) < CTCAE v 3.0 Grade 1.

Exclusion Criteria:

1. Age less than 18 years of age
2. Karnofsky Performance Status less than 60
3. Radiographic or pathologic evidence of metastatic disease (other than pelvic or para-aortic lymph nodes)
4. Prior pelvic radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-04; Primary Completion 2011-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The study will evaluate the feasibility of using helical tomotherapy to deliver IMRT in post-hysterectomy endometrial cancer patients receiving adjuvant radiotherapy. | 1 year from the start of radiation therapy.
  The study will be deemed infeasible if greater than 10% of patients experience one of the following:
  * Patient cannot be given the treatment because her anatomy is such that a dosimetrically satisfactory treatment plan cannot be devised for her.
  * The patient experiences any grade 4 acute toxicity judged to be related to her external radiation treatment.
  * Within 1 year of the start of radiation therapy, the patient develops any grade 4 late toxicity judged to be related to her external radiation treatment.
  * Within 1 year of the start of radiation therapy, the patient develops any in-field pelvic recurrence.
  * Within 1 year of the start of radiation therapy, the patient dies from causes judged to be related to her treatment.

SECONDARY OUTCOMES:
Evaluate incidence of early toxicities | 30 days after last day of radiation therapy
Evaluate incidence of late toxicities | 1 year from the start of radiation therapy
Evaluate local, regional, and distant recurrence rates | 5 years from start of radiation therapy
Evaluate 5-year disease-free and 5-year overall survival rates | 5 years from start of radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Perry W Grigsby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu